CLINICAL TRIAL: NCT03879746
Title: Effect of Tamsulosin on Premature Ejaculation Compared With Paroxetine Hydrochloride
Brief Title: Effect of Tamsulosin on PE Compared With Paroxetine Hydrochloride
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Farrag, Principal Investigator, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: premature ejaculation
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Tamsulosin; Paroxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tamsulosin group (Active Comparator): the first group will include 40 patients treated with daily administration of tamsulosin 0.4 mg
  Interventions: Drug: Tamsulosin
- paroxetine group (Active Comparator): the second group will include 40 patients treated with daily administration of paroxetine 20 mg
  Interventions: Drug: Paroxetine Hydrochloride
- combined group (Active Comparator): the third group will include 40 patients treated with daily administration of tamsulosin 0.4 mg and paroxetine 20 mg
  Interventions: Drug: Tamsulosin; Drug: Paroxetine Hydrochloride
- placrbo group (Placebo Comparator): the fourth group will include 40 patients will be given placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Tamsulosin — drug will be used in treatment of premature ejaculation
  Arms: combined group; tamsulosin group
Drug: Paroxetine Hydrochloride — drug will be used in treatment of premature ejaculation
  Arms: combined group; paroxetine group
Other: placebo — tablets without active substance will be given to patients suffering from premature ejaculation
  Arms: placrbo group

SUMMARY:
A study to compare the effect of tamsulosin versus the effect of paroxetine hydrochloride and the effect of combination of them on PE.

DETAILED DESCRIPTION:
Premature ejaculation is considered the most common male sexual disorder. affecting approximately 4-39 % of men in general community. In 2008, the International Society for Sexual Medicine defined premature ejaculation as a male sexual dysfunction that is characterized by ejaculation that always or nearly always occurs within or before 1 minute of vaginal penetration. Moreover it is associated with presence of distress, frustration, bother, negative personal consequences, depression and the avoidance of sexual intimacy.

Many etiological theories have been included in the pathogenesis of premature ejaculation: neurobiological, psychological, environmental and endocrine factors. So a lot of therapeutic modalities, such as behavioral therapy, selective serotonin reuptake inhibitors (SSRIs), adrenergic alpha 1 antagonists, local anesthetic creams, clomipramine, phosphodiesterase type 5 inhibitors and centrally acting analgesics have been used for the treatment of premature ejaculation.

Previous studies reported that tamsulosin which is alpha blocker agent used as primary therapeutic agent for BPH is effective in the improvement of sexual function. However studies on the effect of tamsulosin on ejaculation reported that tamsulosin had inhibitory effect in the emission phase of ejaculation including decreased ejaculatory volume. So inhibitory effect of tamsulosin on ejaculation may be beneficial to patients suffering from premature ejaculation.

Historically, PE was considered psychological problem and was treated by behavioral treatment and psychotherapy but there is pharmacological studies increase the evidence that PE may be related to decreased serotonergic neurotransmission. So selective serotonin reuptake inhibitors (SSRIs ) such as : paroxetine, fluoxetine, dapoxetine, and sertraline are among the recommended pharmacological treatments for treating PE. But there is no universal agreement on the type, the dose and administration protocol.

So a study is needed to compare the value of combination therapy of both tamsulosin and paroxetine with the value of single therapy of either of them and consider Intravaginal Ejaculatory Latency Time (IELT) and ejaculatory control ability of patients after using tamsulosin and paroxetine.

ELIGIBILITY:
Inclusion Criteria:

* Married, sexually active patients with PE will be included with ages ranging from 20 to 60 years.

Exclusion Criteria:

* Patients suffering from erectile dysfunction, DM, HTN, neurological disorders and psychological disorders.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Premature Ejaculation Diagnostic Tool | 3 months
  Patients will be asked to complete the PEDT ( Premature Ejaculation Diagnostic Tool )
  Cases will be scored as follow :
  * Score of less than or equal 8 indicate no PE .
  * Score of 9 and 10 indicate probable PE .
  * Score of more than or equal 11 indicate PE After about 12 weeks the patients will be reevaluated also by ( PEDT ) and the results will be compared with the pretreatment ones

SECONDARY OUTCOMES:
Intravaginal Ejaculatory Latency Time | 3 months
  Patients will be asked to measure and record (IELT ) during 2 weeks before starting treatment . then they will be asked to measure and record ( IELT ) after each intercourse during and after period of treatment and will be compared with pretreatment measures

IPD SHARING:
Plan to Share IPD: Undecided